CLINICAL TRIAL: NCT00398190
Title: Media Literacy to Prevent Adolescent Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Brian Primack, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 57407
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Smoking Status
Keywords: Smoking; Tobacco use disorder
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Active Comparator): Students receive standard anti-tobacco education
  Interventions: Behavioral: Control
- Media Literacy (Experimental): Students receive media literacy based anti-smoking education
  Interventions: Behavioral: Media Literacy

INTERVENTIONS:
Behavioral: Control — Standard anti-tobacco programming
  Arms: Control
Behavioral: Media Literacy — Anti-smoking media literacy curriculum intervention
  Arms: Media Literacy

SUMMARY:
The purpose of this project is to determine if a 3-session anti-smoking media literacy based intervention is more effective that a standard 3-session anti-smoking media literacy intervention at changing students' intention to smoke, actual smoking behavior, attitudes and norms regarding smoking, and level of media literacy.

DETAILED DESCRIPTION:
Cigarette smoking is the top cause of preventable death and disease in the U.S., and about 90% of those who die from smoking begin as adolescents. Because smoking-related mass media messages (such as episodes of smoking in films and advertisements) significantly increase adolescent smoking, media literacy, defined as analysis and evaluation of mass media messages, presents a promising new framework for development of innovative school-based tobacco control programs. Media literacy may be more effective than standard tobacco education among the populations that are at greatest risk for smoking, such as African-Americans and the socio-economically disadvantaged, and national organizations have called for use of media literacy to reduce smoking. However, anti-smoking media literacy programs have been neither widely implemented nor well-evaluated.

The aims of this project are to determine if a theory-driven, school-based, 3-session anti-smoking media literacy curriculum delivered to 9th grade students can affect clinically relevant factors mediating adolescent smoking according to the widely accepted Theory of Reasoned Action: intention to smoke, smoking behavior, attitude toward smoking, and norms involving smoking. It is hypothesized that, compared with those exposed to a currently accepted school-based smoking prevention program, students exposed to the media literacy program will develop more negative attitudes toward smoking, a more negative sense of smoking norms, less intention to smoke, and less smoking. We also expect that the curriculum will improve smoking media literacy scores as measured by a reliable, valid scale.

Over two years, eight high schools will be recruited to randomize all 9th grade health classrooms to receive either the 3-session media literacy anti-smoking curriculum or a currently accepted anti-smoking program of equivalent length. This recruitment will occur via two prominent community organizations responsible for anti-tobacco programming in 50 local school districts. Experienced health educators will be trained in implementation of both experimental and control curricula. Outcome measures, demographic data, and other important covariates will be collected by a questionnaire given three times: at baseline, immediately post-intervention, and after one year. Questionnaire items are reliable, valid, and pilot-tested. Process evaluation will be conducted to assess implementation fidelity, to confirm or refute the findings of the quantitative assessment, to help explain outcome data, to refine the intervention, and to inform future replications of the curriculum.

Given the substantial nationwide morbidity and mortality due to tobacco use, the role of mass media messages in adolescent initiation of smoking, and the potential power of media literacy as an agent for health behavior change, it is essential to study the utility of media literacy in altering smoking behaviors and antecedents in this age group. If media literacy programs are successful in buffering the impact of mass media on adolescent smoking, similar interventions can be developed to prevent other harmful behaviors related to mass media messages.

ELIGIBILITY:
Inclusion Criteria:

* High school student enrolled in health class at participating schools
* Must be able to use computer interface for submission of data

Exclusion Criteria:

* Child does not wish to participate
* Parent does not wish child to participate
* Less than 13 or more than 18 years old

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1211 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Susceptibility to smoking (Pierce, 1996) | Immediate, Delayed
Current smoking (last 30 days) | Delayed (one year)
Smoking media literacy | Immediate, delayed (one year)

SECONDARY OUTCOMES:
Attitudes toward smoking | Immediate, delayed (one year)
Subjective normative beliefs involving smoking | Immediate, delayed (one year)
Implementation fidelity | Immediate
Feasibility/acceptability of program | Immediate, delayed (one year)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Primack, MD, EdM, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - McKeesport High School, McKeesport, Pennsylvania
  - Carrick High School, Pittsburgh, Pennsylvania
  - Schenley High School, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Primack BA, Gold MA, Land SR, Fine MJ. Association of cigarette smoking and media literacy about smoking among adolescents. J Adolesc Health. 2006 Oct;39(4):465-72. doi: 10.1016/j.jadohealth.2006.05.011. PMID 16982379
- [Background] Primack BA, Gold MA, Switzer GE, Hobbs R, Land SR, Fine MJ. Development and validation of a smoking media literacy scale for adolescents. Arch Pediatr Adolesc Med. 2006 Apr;160(4):369-74. doi: 10.1001/archpedi.160.4.369. PMID 16585481
- [Background] Primack BA, Douglas EL, Land SR, Miller E, Fine MJ. Comparison of media literacy and usual education to prevent tobacco use: a cluster-randomized trial. J Sch Health. 2014 Feb;84(2):106-15. doi: 10.1111/josh.12130. PMID 25099425
- [Background] Primack BA, Fine D, Yang CK, Wickett D, Zickmund S. Adolescents' impressions of antismoking media literacy education: qualitative results from a randomized controlled trial. Health Educ Res. 2009 Aug;24(4):608-21. doi: 10.1093/her/cyn062. Epub 2008 Dec 3. PMID 19052155
- [Background] Primack BA, Hobbs R. Association of various components of media literacy and adolescent smoking. Am J Health Behav. 2009 Mar-Apr;33(2):192-201. doi: 10.5993/ajhb.33.2.8. PMID 18844513